CLINICAL TRIAL: NCT07357428
Title: Connect-One: Early Feasibility Study of Connexus® Brain-Computer Interface (BCI) to Provide Human Connection Through Communication
Brief Title: Connect-One: Early Feasibility Study of Connexus® Brain-Computer Interface (BCI)
Acronym: CONNECT-ONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paradromics (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRT-1014
Record Dates: First submitted 2025-12-23; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Neuromuscular Disease; Stroke; Tetraplegia/Tetraparesis; Cervical Spinal Cord Injury; Dysarthria
Keywords: BCI; ALS; Paradromics; speech; dysarthria; neural injury; progressive neuromuscular disease; stroke; assistive technology; communication device; brain computer interface
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Stroke; Quadriplegia; Dysarthria; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Connect-One (Other)
  Interventions: Device: Connexus Brain-Computer Interface

INTERVENTIONS:
Device: Connexus Brain-Computer Interface — The Connexus Brain Computer Interface is an implantable brain-computer interface.

SUMMARY:
The Connect-One Study is an early feasibility study to obtain preliminary device safety information for the Connexus Brain-Computer Interface (BCI). The Connexus BCI is intended to be used as: (1) an assistive communication device to decode imagined language correlates and speech for patients with impaired communication as a result of severe loss of voluntary motor control; and (2) to provide control of computer devices for individuals with severe loss of voluntary motor control of the upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a progressive neuromuscular disease or a neurological injury.
* Clinical diagnosis of anarthria or severe dysarthria.
* Wheelchair dependent with severely impaired upper limb function.
* Has a reliable method of communication and the ability to read and understand the English language.
* Has a study care partner (e.g. caregiver or multiple caregivers) for the duration of the study.
* Lives within a 4-hour radius of a study site.

Exclusion Criteria:

* Cognitive impairment or psychiatric illness that could impact the ability to comply with study requirements, as determined by the Study Investigator.
* Co-morbidities or an ongoing chronic medical condition that would impair the ability to comply with study requirements.
* The presence of another implanted device, like a pacemaker, deep brain stimulator, or implantable pulse generator.
* Requires, or is expected to require regular MRI scans for on-going medical conditions.
* In the opinion of the Study Investigator, the patient is not an appropriate candidate for the study, for reasons that could place the patient at undue risk or otherwise result in non-compliance with the study requirements.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety: Number of Subjects With Device Related Adverse Events | Up to 12 months post-implant
  Device Related Adverse Events: Number of subjects with device-related adverse events

SECONDARY OUTCOMES:
Long-Term Safety: Number of Subjects With Device Related Adverse Events | Up to 6 years post-implant
  Device Related Adverse Events: Number of subjects with device-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- See also: Paradromics Clinical Study — https://www.paradromics.com/clinical-study